CLINICAL TRIAL: NCT04376489
Title: Novel Use of mHealth Data to Identify States of Vulnerability and Receptivity to JITAIs
Brief Title: Project MARS: Mobile-Assistance for Regulating Smoking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Utah (Other)
Collaborators: University of Michigan (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Wetter, Principal Investigator, University of Utah
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 112287; U01CA229437-01 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-05-06 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Current Smoker; Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking | interventions — cher protein, Drosophila

STUDY DESIGN:
Intervention Model Description: Micro-Randomized Trial (MRT) in the development of data-driven behavioral interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief cognitive/behavioral strategies (Experimental)
  Interventions: Behavioral: Messages (participants experiencing negative affect & cigarettes are available); Behavioral: Messages (participants not experiencing negative affect & cigarettes are available); Behavioral: Messages (participants experiencing negative affect & cigarettes are not available); Behavioral: Messages (participants not experiencing negative affect & cigarettes are not available)
- Effortful self-regulatory activities (Experimental)
  Interventions: Behavioral: Moodsurf; Behavioral: Meditate; Behavioral: Joy; Behavioral: Imagine; Behavioral: Notice
- No activities (No Intervention)

INTERVENTIONS:
Behavioral: Messages (participants experiencing negative affect & cigarettes are available) — Participants receive messages tailored for situations when they experiencing negative affect & cigarettes are available.
  Arms: Brief cognitive/behavioral strategies
Behavioral: Messages (participants not experiencing negative affect & cigarettes are available) — Participants receive messages tailored for situations when they cigarettes are available.
  Arms: Brief cognitive/behavioral strategies
Behavioral: Messages (participants experiencing negative affect & cigarettes are not available) — Participants receive messages tailored for situations when they experiencing negative affect.
  Arms: Brief cognitive/behavioral strategies
Behavioral: Messages (participants not experiencing negative affect & cigarettes are not available) — Generic messages for situations when participants are neither experiencing negative affect nor cigarettes are available.
  Arms: Brief cognitive/behavioral strategies
Behavioral: Moodsurf — Smart phone app that teaches participants a mindfulness-based technique in which participant "surf" the mood.
  Arms: Effortful self-regulatory activities
Behavioral: Meditate — Smart phone app that teaches participants a mindfulness-based meditation designed for smoking cessation.
  Arms: Effortful self-regulatory activities
Behavioral: Joy — Smart phone app that teaches participants to practice breathing exercise.
  Arms: Effortful self-regulatory activities
Behavioral: Imagine — Smart phone app that teaches participants to use their imagination to explore and manage their thoughts and feelings.
  Arms: Effortful self-regulatory activities
Behavioral: Notice — Smart phone app that teaches participants to accept their thoughts and feelings.
  Arms: Effortful self-regulatory activities

SUMMARY:
This study aims to identify states of vulnerability for lapse, identify states of receptivity for engaging in self-regulatory activities, and investigate approaches to capitalize on states of vulnerability and receptivity to deliver real-time self-regulation prompts among smokers.

DETAILED DESCRIPTION:
Aim 1: Identify states of vulnerability for lapse: Self-reported and sensor-based measures will be used to identify empirically-based and theoretically-grounded features across multiple time scales that are most predictive of lapse. Operationalizing vulnerability in terms of the predicted level of risk for lapse, the investigators hypothesize that (H1) current vulnerability is represented by current and/or recent high negative emotions, low positive emotions, high craving, low self-efficacy, low self-regulatory capacity (SRC), and risky context (e.g., specific locations, such as a bar; cigarettes available; others smoking).

Aim 2: Identify states of receptivity for engaging in self-regulatory activities: Self-reported and sensor-based measures will be used to identify empirically-based and theoretically-grounded features across multiple time scales that are most predictive of engagement (i.e., usage of self-regulatory activities). Operationalizing receptivity in terms of the predicted likelihood of engagement, the investigators hypothesize that (H2) current receptivity is represented by high positive activating emotions (e.g., happy, grateful), low negative deactivating emotions (e.g., sad, boredom), low craving, high self-efficacy, high SRC, and low risk contexts (e.g., specific locations, such as home).

Aim 3: Investigate approaches to capitalize on states of vulnerability and receptivity to deliver real-time self-regulation prompts. Investigate whether, what type, and under what conditions (e.g., current state of vulnerability and/or receptivity) a prompt to engage the individual in self-regulatory activities increases engagement, hence reduces vulnerability.

The proposed research will help build a comprehensive conceptual, technical, and empirical foundation necessary to develop effective Just-in-Time-Adaptive-Interventions (JITAIs) based on dynamic models of vulnerability and receptivity. In the micro-randomized trial (MRT), Ecological momentary assessments (EMAs) are administered before and after JITAIs with items that are designed to measure different indices that may be related to participants' engagement of the JITAIs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current smoker with an average of at least 3 cigarettes/day
* Motivated to quit within the next 30 days
* Valid home address
* Functioning telephone number
* Can speak, read, and write in English
* At least marginal health literacy (as determined by 45 or greater on REALM literacy test)

Exclusion Criteria:

* Contraindication for nicotine patch
* Current use of tobacco cessation medications or other aids (i.e. buproprion)
* Pregnancy or lactation (as self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Biochemically Verified Smoking Abstinence | Post-quit date - 6-month follow-up
  Smoking abstinence will be completed via self-reported status from participants which are biochemically verified by either expired carbon monoxide via a breathalyzer or a cotinine sample as needed if a participant is unable to attend a visit in-person.

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, PhD, Principal Investigator — University of Utah; Inbal Nahum-Shani, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA). Before sharing data, data will be stripped of all personal identifiers and all identifying codes. Data will be deemed either sensitive or low-risk, based on our characterization of the possibility of deductive disclosure. Request for sensitive data will be vetted through an assessment of both the requestor's credentials and potential risks. Note that our risk analysis will be based on a joint consideration of the total risk based on all data products requested.
Supporting Information: Study Protocol, SAP
Time Frame: The PIs and the research team will work to make the data available in a reasonable amount of time after its collection and following the acceptance for publication of the main findings. Rules for maintaining and distributing data of the University of Utah, the University of Michigan, and the NIH will be followed.